CLINICAL TRIAL: NCT03199625
Title: Different Neural Circuit Mechanisms Between Cognitive Therapy and Behavior Therapy for Patients With Panic Disorder: a Dynamic Research
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Chun Wang, Nanjing Brain hospital, Nanjing Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 81571344
Record Dates: First submitted 2017-06-20; First posted 2017-06-27 (Actual); Last update posted 2017-06-27 (Actual); Status verified 2016-12

CONDITIONS: Panic Disorder
Keywords: cognitive-behavior therapy; magnetic resonance imaging; Panic Disorder
MeSH Terms: conditions — Panic Disorder | interventions — Cognitive Behavioral Therapy; Behavior Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- Cognitive Therapy group (Experimental): treatment with Cognitive Therapy
  Interventions: Behavioral: Cognitive therapy
- Behavior Therapy group (Experimental): treatment with Behavior Therapy
  Interventions: Behavioral: Behavior therapy
- SSRI antidepressants (Active Comparator): treatment by SSRI antidepressant
  Interventions: Drug: SSRI antidepressants

INTERVENTIONS:
Behavioral: Cognitive therapy
  Other Names: cognitive therapy(CT)
  Arms: Cognitive Therapy group
Behavioral: Behavior therapy
  Other Names: Behavior therapy(BT)
  Arms: Behavior Therapy group
Drug: SSRI antidepressants
  Arms: SSRI antidepressants

SUMMARY:
Cognitive behavioral therapy (CBT), which includes cognitive therapy (CT) and behavioral therapy (BT), is the first-line treatment for patients with panic disorder (PD). However, the neural mechanism of CBT is unknown. The exploration of mechanism is of great significance for clinical strategy formulation. This study is proposed on the basis of our early PD and CBT neuroimaging studies, adopt the design of prospective randomized controlled intervention study, set up three time points: before the treatment（week 0）, the initial treatment (week 4th), the plateau treatment (week 28th). With normal subjects as black control and antidepressant therapy as intervention comparison, this study set up CT and BT two intervention groups, respectively collect all the participants'symptomatological, psychological, cognitive function and brain imaging data (3D,DTI, fMRI in resting and tasks states) at week 0, week 4th and week 28th. This study is based on the advanced analysis methods we applied in the early study,including BOLD-fMRI, DTI, topological characteristics analysis of the whole brain network and Granger causality test etc. It is from the point of multiple levels(brain regions, circuits, whole brain), multimodal (structure, function) to comprehensively analysis the role of CT and BT for the function and structure of brain regions, circuits (mood regulating circuit and cognitive control network for emotion processing) and whole brain in patients with PD. Totally, we explore the target area, path and mechanism of CBT for emotion processing neural circuits in patients with PD, and combined with the clinical data we preliminarily explore the imaging biomarkers of different intervention methods which may predict therapeutic effect.

ELIGIBILITY:
Inclusion Criteria:

* meet DSM-5 and Mini-international neuropsychiatric interview (MINI) Chinese version panic disorder diagnosis;
* the age of 20-50 years old;
* Right handedness;
* patients to participate voluntarily, with the consent of their families, signed informed consent book.

Exclusion Criteria:

* neurological diseases or other mental illnesses;
* serious physical illness (e.g. heart, lung, liver, kidney or blood system disease);
* treatment by psychotropic medications,psychological treatment, electroconvulsive therapy or physical therapy within 3 months prior to the start of the trial;
* with contraindication for MRI
* pregnancy and lactation.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 96 (Estimated)
Dates: Start 2016-01; Primary Completion 2018-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Hamilton Anxiety Scale behavior therapy for patients with panic disorder: a dynamic research | an expected average of 6 months
  The 14-item version of the Hamilton Rating Scale for Anxiety (HAMA; Hamilton, 1959) will be used for measuring severity of depressive symptoms. Minimum and maximum possible values are respectively 0 and 56. Lower scores show more mild anxiety.
Magnetic Resonance Imaging | Time Frame: an expected average of 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Chun Wang, doctor, Principal Investigator — Nanjing Medical University
Locations (1):
- Nanjing Brain Hospital, Nanjing, Jiangsu, China